CLINICAL TRIAL: NCT06024603
Title: Individualized Treatments in Adults With Relapsed/Refractory Cancers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Florida International University (Other); Community Foundation of Broward (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5Y22
Record Dates: First submitted 2023-07-28; First posted 2023-09-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Refractory Cancer; Relapsed Cancer
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug Sensitivity Testing (Experimental): The results of the DST and genomic screening will be used to inform treating physician about participant-specific drug sensitivity or resistance guiding best therapy choices. The physician will decide which treatment will be most appropriate for each case. All participants will need to be consented separately for any subsequent investigational treatment if no standard treatment options are available.
  Interventions: Diagnostic Test: Drug Sensitivity Test (DST)

INTERVENTIONS:
Diagnostic Test: Drug Sensitivity Test (DST) — Refractory cancer tissue will be collected from participants and subjected to single-drug testing while DNA is simultaneously sent for targeted gene sequencing. Drug sensitivity scores from the tests will become available for a final list of therapeutic options ranked best in order of preference together with suggested doses and schedules.

SUMMARY:
A personalized cancer medicine approach would address therapy resistance, cancer metastasis, and limited options after standard of care is exhausted in advanced cancer participants. This approach may reduce the barriers to approved therapeutic assignment currently limited to a particular cancer type or patient demographic.

DETAILED DESCRIPTION:
Treatment itself will not be given as part of this trial. The results of the drug sensitivity test (DST) and genomic screening will be used to inform treating physician about participant-specific drug sensitivity or resistance guiding best therapy choices. The physician will decide the most appropriate treatment for each case, with the option to add one or more personalized (assay-guided) drug(s) from the investigational platform. All participants will need to be consented separately for any subsequent investigational treatment if no standard treatment options are available.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older at the time of enrollment on this study of any gender, race, or ethnicity.
* Patients with suspected or confirmed diagnosis of recurrent or refractory cancer with no curative treatment options.
* Participants who have undergone at least two lines of previous therapy.
* Participants who are scheduled for or have recently had biopsy or tumor excised (solid tumors) or bone marrow aspirate (blood cancers) or who have scheduled or recently had paracentesis or thoracentesis performed.
* Participants willing to have a blood draw or buccal swab done for the purposes of genetic testing.
* Participants willing to sign informed consent.

Exclusion Criteria:

* Participants who do not have malignant tissue available and accessible.
* Participants for whom the amount of excised malignant tissue is not sufficient for the ex vivo drug testing and/or genetic profiling.
* Participants with newly diagnosed tumors and tumors that have high (>90%) cure rate with safe standard therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment recommendation feasibility | Up to 4 weeks post-treatment
  Primary objective is to determine feasibility of providing treatment recommendations to relapsed and refractory adult cancer patients based on ex vivo drug sensitivity testing (DST). Feasibility will be demonstrated if it is possible to recommend treatment within 4 weeks in at least 22 of 36 participants (62.5%).
Treatment recommendation feasibility | Up to 4 weeks post-treatment
  Primary objective is to determine feasibility of providing treatment recommendations to relapsed and refractory adult cancer patients based on genomic profiling. Feasibility will be demonstrated if it is possible to recommend treatment within 4 weeks in at least 22 of 36 participants (62.5%).

SECONDARY OUTCOMES:
Treatment responsiveness | Up tp 1 year post-treatment
  Treatment responsiveness will be measured by comparing individual outcomes of adult participants with relapsed and refractory cancers treated with DST-guided therapy to non-DST guided (conventional) therapy. To address this goal, the overall response rate will be calculated. A responder to the treatment will be defined as any patient who achieves a best response of "partial response" or "complete response" during the study period. Evaluable patients who demonstrate a complete or partial response confirmed by physician's review will be considered a responder. All other evaluable patients will be considered non- responder. Outcomes will be observed during treatment and follow-up for one year post-treatment or until disease progression, death, or withdrawal, whichever occurs first.
Progression-free survival | Up tp 1 year post-treatment
  Progression-free survival will be measured by comparing individual outcomes of participants with relapsed and refractory cancers treated with DST-guided therapy to non-DST guided (conventional) therapy. DFS will be defined as time from start of treatment to even (treatment failure, relapse, second malignancy, death) or last follow-up for those who are event-free. Outcomes will be observed during treatment and follow-up for one year post-treatment or until disease progression, death, or withdrawal, whichever occurs first.
Progression-free survival ratio | Up to 1 year post-treatment
  We will assess changes in progression-free survival from each patient's previous treatment versus their progression-free survival from the treatment assigned during the trial. Assessments will be made both in the DST-guided cohort and the non-DST-guided (conventional) cohort. Analysis will include both the raw ratio as well as the number of incidences of 30% improved PFS on trial versus previous regimen (PFS2/PFS1 > 1.3x).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Manrique-Succar, MD, Principal Investigator — Lerner College of Medicine, Cleveland Clinic Florida; Diana Azzam, PhD, Principal Investigator — Robert Stempel College of Public Health and Social Work, Florida International University
Locations (2):
- United States (2):
  - Florida International University, Miami, Florida
  - Lerner College of Medicine, Cleveland Clinic Florida, Weston, Florida